CLINICAL TRIAL: NCT05549232
Title: A Single Center, Pilot Clinical Investigation of Surgical Bleeding in Burn Patients, and Chronically Transfused Patients With Haematologic Malignancies, Who Are Transfused With Hypoxic Red Blood Cells Manufactured With Hemanext ONE System
Brief Title: Hypoxic Red Blood Cells for Burns and Hematological Malignancies at Haukeland University Hospital
Status: Completed | Type: Observational
Sponsor: Hemanext (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-CLIN-0012
Record Dates: First submitted 2022-08-29; First posted 2022-09-22 (Actual); Results first posted 2025-05-18 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Hematologic Neoplasms; Burns
Keywords: Transfusion; Red Blood Cells; Hypoxic
MeSH Terms: conditions — Hematologic Neoplasms; Burns; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Hematologic Malignancies: Subjects requiring chronic transfusions with red blood cells for treatment of a hematologic malignancy will receive 1 transfusion with 2 units of hypoxic red blood cells manufactured with the Hemanext ONE device. The subjects will be monitored for all adverse events from Informed Consent through Day 28 or the subsequent standard of care transfusion, whichever occurs first.
  Interventions: Device: Hypoxic Red Blood Cells
- Acute Burn: Subjects requiring transfusion with red blood cells during the excision procedure after an acute burn will receive 2 units of hypoxic red blood cells manufactured with the Hemanext ONE device. As the excision treatments require transfusion of more than 2 units of red blood cells, the first 2 units transfused during the procedure will be hypoxic red blood cells. The subjects will be monitored for all adverse events through Day 28.
  Interventions: Device: Hypoxic Red Blood Cells

INTERVENTIONS:
Device: Hypoxic Red Blood Cells — Hypoxic Red Blood Cells manufactured with the Hemanext ONE device- CPD/PAGGSM Red Blood Cells, Leukocytes Reduced, and O2/CO2 Reduced

SUMMARY:
The overall objective of this study is to collect preliminary safety data on the transfusion of hypoxic RBCs, manufactured with the Hemanext ONE device, in patients with burns and patients with hematological malignancies. The Hemanext ONE device received CE mark in April 2021.

DETAILED DESCRIPTION:
The primary objective is to assess hypoxic RBCs safety and tolerance assessment up to 24 hours following the transfusion initiation and overall up to 7 days (+/- 1 day) after the transfusion episode (single transfusion course).

Secondary objectives include the following.

1. Assessment of pre and post transfusion hemoglobin levels
2. Assessment of hemoglobin level before the following transfusion, if applicable
3. Assessment of AEs occurrence:

   i. Up to 7 days (+/- 1 day) post transfusion, in comparison with historical control (including but not limited to infection, deep vein thrombosis, acute respiratory distress syndrome, transfusion-related acute lung injury, transfusion associated circulatory overload, anaphylactic shock, acute hemolytic transfusion reaction).

   ii. Up to the subsequent transfusion episode or up to 28 days (+/- 1 day) after the initial transfusion, whichever comes first.

   iii. From enrollment, up to their subsequent transfusion or 28 days (+/- 1 day) post transfusion, whichever comes first, through the assessment of patient's diary.
4. Assessment of the vital signs during and up to 15 minutes after the transfusion.

ELIGIBILITY:
Inclusion Criteria:

A. Hematological malignancies patients group:

1. Male or female patients at least 18 years of age
2. Patients expected to require > 2 units of red blood cells in a single transfusion event
3. Patients who have the capacity to consent to participate and are willing to comply with the study procedures.
4. Patients identified by a Transfusion hemoglobin trigger of less than 9 g/dL
5. Patients with a documented diagnosis of leukemia, myelomatosis or MDS requiring chronic transfusions

B. Burn patients group:

1. Male or female patients at least 18 years of age
2. Patients who have the capacity to consent by themselves to participate to the clinical investigation
3. Smaller burn patients, hospitalized with a Total Body Surface Area (TBSA%) burn ≥ 10% and ≤ 50%
4. Patients expected to require > 2 unit of red blood cells in a single transfusion event

Exclusion Criteria:

A. Both patients groups

1. Patients with any positive antibody screening test
2. Patients for whom consent has not been obtained
3. Patients with a known hemolytic anemia (congenital or acquired)
4. Patients < 18 years old
5. Patients with a known or suspected pregnancy
6. Patients with a history of major transfusion reactions
7. Patients whom the Investigator deems clinical trial participation is not in their best interest.

B. Burn patients specific exclusion criteria :

1. Patients who do not have the capacity to consent by themselves to participate to the clinical investigation
2. Patients hospitalized with a Total body surface area (TBSA%) burn more than 50%
3. Patients with combined trauma in need of blood transfusions for treatment other than the burn excision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 acute burn patients and 10 patients with hematological malignancies, who require transfusion of red cells concentrates and who fulfill all eligibility criteria will be enrolled in this clinical investigation at Haukeland University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoshida T, Prudent M, D'alessandro A. Red blood cell storage lesion: causes and potential clinical consequences. Blood Transfus. 2019 Jan;17(1):27-52. doi: 10.2450/2019.0217-18. PMID 30653459
- [Background] Williams AT, Jani VP, Nemkov T, Lucas A, Yoshida T, Dunham A, D'Alessandro A, Cabrales P. Transfusion of Anaerobically or Conventionally Stored Blood After Hemorrhagic Shock. Shock. 2020 Mar;53(3):352-362. doi: 10.1097/SHK.0000000000001386. PMID 31478989
- [Background] D'Alessandro A, Yoshida T, Nestheide S, Nemkov T, Stocker S, Stefanoni D, Mohmoud F, Rugg N, Dunham A, Cancelas JA. Hypoxic storage of red blood cells improves metabolism and post-transfusion recovery. Transfusion. 2020 Apr;60(4):786-798. doi: 10.1111/trf.15730. Epub 2020 Feb 27. PMID 32104927

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hematologic Malignancies | Acute Burn
Started | 10 | 12
Completed | 9 | 10
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hematologic Malignancies | Acute Burn | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 10 | 12
  >=65 years | 8 | 2 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.0 (16.41) | 49.6 (19.46) | 59.8 (21.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 8 | 10 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 11 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Norway | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event (All Types/Grades) Within a Time Frame up to 24 Hours Following the Transfusion.
Description: The type and the grade of each adverse event will be categorized according to:
  * Association for the Advancement of Blood and Biotherapies (AABB) technical manual, 20th edition (2020)
  * Biomedical Excellence for Safer Transfusion (BEST) Collaborative review - Lancet 2016; 388: 2825-36
  * Local AEs database (for reference)
  * ISO 14155-2020 definitions
Time Frame: 24 hours
Population: Participants in the Safety analysis set who experienced an adverse event (all types/grades) within a time frame up to 24 hours following transfusion. Participants who did not receive a transfusion were not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Hematologic Malignancies | Acute Burn
Number analyzed (Participants) | 10 | 10
Participants | 2 | 3

2. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE) (All Types/Grades) Overall up to 7 Days (+/-1 Day) After the Transfusion.
Description: as for outcome 1
Time Frame: 7 days (+/-1 day)
Population: Participants in the Safety analysis set. Participants who did not receive a transfusion were not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Hematologic Malignancies | Acute Burn
Number analyzed (Participants) | 10 | 10
Participants | 4 | 7

3. Secondary Outcome: Evolution of the Hemoglobin Level Before and After the Transfusion.
Description: The difference in measured hemoglobin (grams/dL) between pre-transfusion and up to 30 minutes post-transfusion.
Time Frame: pre-transfusion to up to 30 minutes post-transfusion
Population: Safety analysis set. Participants who did not receive a transfusion were not included in the analysis
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Hematologic Malignancies | Acute Burn
Number analyzed (Participants) | 10 | 10
g/dL | 1.20 (0.494) | 0.25 (0.981)

4. Secondary Outcome: Calculation of the Hemoglobin Increment After Transfusion Corrected for Patient Blood Volume and Hemoglobin Dose
Description: The hemoglobin increment from each transfusion will be determined by calculating the difference between the subject's post-transfusion and pre-transfusion hemoglobin (g/dL). It will then be corrected for estimated subject blood volume and the amount of Hb transfused.
  The following equation used for the hemoglobin increment calculation:
  HgB Increment = (Subject's HgB level post-transfusion - Subject's HgB pre-transfusion)/ (total HgB transfused x Subject's BloodVolume)
  Equations for calculating the hemoglobin increment may be found in the following publication: Wendelbo Ø, Opheim EN, Hervig T, Felli Lunde TH, Bruserud Ø, Mollnes TE, Reikvam H. Cytokine profiling and post-transfusion haemoglobin increment in patients with haematological diseases. Vox Sang. 2018 Oct;113(7):657-668. doi: 10.1111/vox.12703. Epub 2018 Aug 29. PMID: 30159896.
Time Frame: 28 days
Population: Outcome not analyzed. The reason for this change is that it was not possible to calculate the hemoglobin increment from the collected data. Patient HgB results were collected pre and post transfusion. However, total HgB transfused (i.e. how much HgB was present in RBC units) was not assessed. This missing variable is required to complete the HgB Increment calculation, which prevented us from completing the calculation in order to report adjusted hemoglobin increment.
Arm/Group | Hematologic Malignancies | Acute Burn
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Comparison of the Hemoglobin Level Before the Index Transfusion to That Prior to the Subsequent Transfusion
Description: The difference in measured hemoglobin (grams/dL) between the pre-transfusion hemoglobin level for the study transfusion and the pre-transfusion hemoglobin level for the next scheduled transfusion.
Time Frame: 28 days
Population: Safety analysis set. Participants who did not receive a transfusion were not included in the analysis.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Hematologic Malignancies | Acute Burn
Number analyzed (Participants) | 10 | 10
g/dL | 0.21 (1.177) | 0.84 (2.065)

6. Secondary Outcome: Evaluation of AEs From Enrollment, up to Prior to the Subsequent Transfusion or up to Day 28, Whichever Occurs First
Description: Number of AEs that occur from enrollment, up to prior to the subsequent transfusion or up to Day 28, whichever occurs first
Time Frame: 28 days
Population: Safety analysis set. Participants who did not receive a transfusion were not included in the analysis.
Measure: Number; unit: adverse event
Arm/Group | Hematologic Malignancies | Acute Burn
Number analyzed (Participants) | 10 | 10
adverse event | 4 | 7

7. Secondary Outcome: Evaluation of Subject's Blood Pressure Over the Course of the Transfusion and up to 15 Minutes Post-transfusion
Description: Change in blood pressure (systolic; mmHg) from baseline up to 15 minutes post-transfusion.
Time Frame: baseline up to 15 minutes post-transfusion.
Population: Safety analysis set. Participants who did not receive a transfusion were not included in the analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Hematologic Malignancies | Acute Burn
Number analyzed (Participants) | 10 | 10
mmHg | -4.56 (6.521) | -3.40 (23.996)

8. Secondary Outcome: Evaluation of Subject's Blood Pressure Over the Course of the Transfusion and up to 15 Minutes Post-transfusion
Description: Change in blood pressure (diastolic; mmHg) from baseline up to 15 minutes post-transfusion.
Time Frame: baseline up to 15 minutes post-transfusion.
Population: Safety analysis set. Participants who did not receive a transfusion were not included in the analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Hematologic Malignancies | Acute Burn
Number analyzed (Participants) | 10 | 10
mmHg | -0.44 (7.333) | 1.90 (9.219)

9. Secondary Outcome: Evaluation of Subject's Respiratory Rate Over the Course of the Transfusion and up to 15 Minutes Post-transfusion
Description: Change in respiratory rate (breaths per minute) from baseline to up to 15 minutes post-transfusion.
Time Frame: baseline to up to 15 minutes post-transfusion
Population: Safety analysis set. Participants who did not receive a transfusion were not included in the analysis.
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Hematologic Malignancies | Acute Burn
Number analyzed (Participants) | 10 | 10
breaths/min | 0.00 (2.062) | -1.10 (2.846)

10. Secondary Outcome: Evaluation of Subject's SO2 Level Over the Course of the Transfusion and up to 15 Minutes Post-transfusion
Description: Change in the amount of oxygen in the body (% S02 level), measured with a pulse oximeter, from baseline to up to 15 minutes post-transfusion.
Time Frame: baseline to up to 15 minutes post-transfusion
Population: Safety analysis set. Participants who did not receive a transfusion were not included in in analysis.
Measure: Mean (Standard Deviation); unit: % O2 saturation
Arm/Group | Hematologic Malignancies | Acute Burn
Number analyzed (Participants) | 10 | 10
% O2 saturation | 0.22 (1.856) | 0.00 (1.633)

11. Secondary Outcome: Evaluation of Subject's Pulse Over the Course of the Transfusion and up to 15 Minutes Post-transfusion
Description: Change in heart rate (beats per minute) from baseline to up to 15 minutes post-transfusion
Time Frame: baseline to up to 15 minutes post-transfusion
Population: Safety analysis set. Participants who did not receive a transfusion were not included in analysis.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Hematologic Malignancies | Acute Burn
Number analyzed (Participants) | 10 | 10
beats/min | -3.33 (6.144) | 5.40 (16.263)

ADVERSE EVENTS:
Time Frame: Adverse Events reported up to 28 days post-transfusion, or up to subsequent transfusion episode, whichever comes first
Description: The type and the grade of each adverse event were categorized according to:
  * Association for the Advancement of Blood and Biotherapies (AABB) technical manual, 20th edition (2020)
  * Biomedical Excellence for Safer Transfusion (BEST) Collaborative review - Lancet 2016; 388: 2825-36
  * Local AEs database (for reference)
  * ISO 14155-2020 definitions
Arm/Group | Hematologic Malignancies | Acute Burn
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/12
Other Adverse Events (participants affected / at risk) | 4/10 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematologic Malignancies (N=10) | Acute Burn (N=12)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematologic Malignancies (N=10) | Acute Burn (N=12)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Catheter site extravasation (General disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Spinal operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall provide Sponsor with a copy of the papers, abstracts or presentations not less than thirty (30) days prior to submission to a scientific journal or presentation at scientific meetings. Sponsor shall have thirty (30) days to review the proposed publication. Sponsor may comment upon, but may not make any editorial changes to, the results and conclusions set forth in the papers unless Confidential Information is identified and must be deleted.

DOCUMENTS (2):
  • Study Protocol (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/32/NCT05549232/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT05549232/SAP_001.pdf